CLINICAL TRIAL: NCT03810378
Title: Contrasting Ketogenic and Mediterranean Diets in Individuals With Type 2 Diabetes and Prediabetes: The Keto-Med Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Christopher Gardner, Professor of Medicine, Stanford University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 49218
Record Dates: First submitted 2019-01-09; First posted 2019-01-18 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Diabetes Mellitus, Type 2; PreDiabetes
Keywords: Ketogenic diet; Mediterranean diet; Diabetes; Prediabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Prediabetic State; Diabetes Mellitus | interventions — Diet, Mediterranean

STUDY DESIGN:
Intervention Model Description: 40 adults will be randomized in cross-over design to a Ketogenic or Mediterranean diet for 12 weeks each (no washout) with a 1 month follow-up at the end of the second phase.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mediterranean Diet (Med-Plus) (Experimental): Participants will follow a Mediterranean-type diet (Med-Plus) for 12 weeks. This diet will maximize the intake of vegetables, legumes, fruits and nuts, whole intact grains/cereals and fish; and minimize the intake of meat, poultry, and dairy. It will exclude added sugars and refined grains.
  Interventions: Behavioral: Mediterranean Diet (Med-Plus)
- Well-Formulated Ketogenic Diet (WFKD) (Experimental): Participants will follow a Well-Formulated Ketogenic Diet (WFKD) for 12 weeks. This diet will maximize the intake of non-processed beef, pork, and poultry (preferably organic/grass-fed), fish, heavy cream, low-lactose, high-fat cheeses, animal fats, oils (avocado, coconut, or other nut oils), non-starchy (above ground) vegetables and limited amounts of some fruits (berries). It will exclude legumes, grains, sugars, starchy (below ground) vegetables, most fruits, and polyunsaturated oils (soy, sunflower, peanut, cottonseed, canola, etc.). It will aim for an intake of 20 g of carbohydrates/day at start, with the goal to have no more than 50 grams/day to maintain ketosis.
  Interventions: Behavioral: Well-Formulated Ketogenic Diet (WFKD)

INTERVENTIONS:
Behavioral: Mediterranean Diet (Med-Plus) — Participants will follow the Med-Plus diet for 12 weeks, then switch to the alternate diet for another 12 weeks (no washout period).
  Arms: Mediterranean Diet (Med-Plus)
Behavioral: Well-Formulated Ketogenic Diet (WFKD) — Participants will follow the WFKD diet for 12 weeks, then switch to the alternate diet for another 12 weeks (no washout period).
  Arms: Well-Formulated Ketogenic Diet (WFKD)

SUMMARY:
The objective of this study is to compare two metabolically distinct diets, WFKD vs Med-Plus, in order to examine the potential benefits, and unintended consequences, of going beyond a focus on maximally avoiding added sugars and refined grains, to also avoiding legumes, fruits, and whole grains.

DETAILED DESCRIPTION:
The proposed randomized clinical trial will investigate differential population-specific effects of two low-carbohydrate (low-carb) diet patterns, addressing a gap in the evidence base in this area that will lead to 1) improved treatment strategies for common adverse clinical conditions, 2) improved health for these individuals, and 3) long-term decreases in health care costs. This impactful research will advance the field of personalized and precision medicine.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18
* Diagnosed with type 2 diabetes mellitus, OR prediabetes (defined as HbA1c </= 5.7% OR Fasting Glucose of >100 mg/dL)

Identify exclusion criteria.

* Weight < 110 lb
* BMI > 40
* LDL-C >190 mg/dL
* Blood pressure: SBP > 160 mmHg OR DBP: > 90 mmHg

Exclusion Criteria:

* Weight < 110 lb
* BMI ≥ 40
* LDL-C >190 mg/dL
* Systolic blood pressure (SBP) > 160 mmHg OR Diastolic blood pressure (DBP) > 90 mmHg
* Diagnosed with type 1 diabetes or history of ketoacidosis
* Uncontrolled and untreated diabetes (by discretion of study physician)
* Active cardiovascular disease (in past year with myocardial infarction, coronary stent or bypass surgery)
* Kidney disease (eGFR less than 50 mL/min per 1.73 m2)
* Liver disease (liver transaminase higher than 3 times the normal range for the laboratory)
* Symptomatic gallstones
* History of bariatric surgery
* Anemia
* Taking any of the following medications in past 3 months: SGLT-2 inhibitors, GLP-1 receptor agonist, Insulin, Amylin analog, Alpha-glucosidase inhibitor, Dopamine agonist, Bile acid sequestrant.
* Taking any medications for weight loss
* History of active cancer in the past 3 years except for squamous or basal cell carcinomas of the skin that have been medically managed by local excision
* Unstable dietary history as defined by major changes in diet during the previous month, where the subject has eliminated or significantly increased a major food group in the diet.
* Recent history of chronic excessive alcohol consumption defined as more than five 1.5-ounce servings of 80 proof distilled spirits, five 12-ounce servings of beer or five 5-ounce servings of wine per day; or > 14 drinks/week.
* Women: Pregnant currently or planning to become pregnant during the course of the study, and/or breastfeeding
* Regular/frequent use of smoking or chewing tobacco, e-cigarettes, cigars or other nicotine-containing products
* Regular use of prescription opiate pain medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2019-06-05 (Actual); Primary Completion 2020-12-04 (Actual); Study Completion 2020-12-06 (Actual)

PRIMARY OUTCOMES:
Hemoglobin A1c (HbA1c) | Baseline and 12 weeks
  Change from baseline in HbA1c at 12 weeks of each phase

SECONDARY OUTCOMES:
Microbiota composition | Baseline and 12 weeks
  Change from baseline in alpha diversity at 12 weeks of each phase. We will be using number of observed sequence variants ("species") determined by standard 16S rRNA amplicon sequencing (V3-V5 region followed by DADA2 to define error-corrected sequence variants) as our primary metric of alpha diversity. Higher alpha diversity is better. The units are the # of sequence variants.
Microbiota function | Baseline and 12 weeks
  Change from baseline in composite of short-chain fatty acids (SCFA) concentration (ug/g stool: acetate + propionate + butyrate) at 12 weeks of each phase.
LDL Cholesterol | Baseline and12 weeks
  Change from baseline in LDL cholesterol at 12 weeks of each phase.
HDL Cholesterol | Baseline and 12 weeks
  Change from baseline in HDL cholesterol at 12 weeks of each phase.
Triglycerides | Baseline and 12 weeks
  Change from baseline in triglycerides at 12 weeks of each phase.
Fasting insulin | Baseline and 12 weeks
  Change from baseline in fasting insulin at 12 weeks of each phase.
Blood pressure | Baseline and 12 weeks
  Change from baseline in blood pressure at 12 weeks of each phase.

OTHER OUTCOMES:
Satisfaction with WFKD and Med-Plus diets | Baseline and 12 weeks
  Average satisfaction level with meals at 12 weeks of each phase (WFKD compared to Med-Plus phase) using a 5-point Likert scale (1=not at all satisfied; 2=slightly satisfied; 3=moderately satisfied; 4=very satisfied; 5=extremely satisfied).
Adherence to diet protocols | Baseline and 12 weeks
  Adherence to diet protocols 12 weeks of each phase in subjects with Diabetes compared to subjects with prediabetes, according to 3-day food records.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Gardner, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gardner CD, Landry MJ, Perelman D, Petlura C, Durand LR, Aronica L, Crimarco A, Cunanan KM, Chang A, Dant CC, Robinson JL, Kim SH. Effect of a ketogenic diet versus Mediterranean diet on glycated hemoglobin in individuals with prediabetes and type 2 diabetes mellitus: The interventional Keto-Med randomized crossover trial. Am J Clin Nutr. 2022 Sep 2;116(3):640-652. doi: 10.1093/ajcn/nqac154. PMID 35641199
- [Derived] Landry MJ, Crimarco A, Perelman D, Durand LR, Petlura C, Aronica L, Robinson JL, Kim SH, Gardner CD. Adherence to Ketogenic and Mediterranean Study Diets in a Crossover Trial: The Keto-Med Randomized Trial. Nutrients. 2021 Mar 17;13(3):967. doi: 10.3390/nu13030967. PMID 33802709
- See also: Study description and summary of results — https://med.stanford.edu/nutrition/research/completed-studies/KETOMEDstudy.html

DOCUMENTS (1):
  • Statistical Analysis Plan (2020-12-18): https://cdn.clinicaltrials.gov/large-docs/78/NCT03810378/SAP_000.pdf